CLINICAL TRIAL: NCT06506058
Title: Vestibular and Cortical Contributions to Transitions in Freezing of Gait in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NEUR-2024-33325
Record Dates: First submitted 2024-06-13; First posted 2024-07-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: The study will use a cross-sectional design to examine the effects of group (PD with FOG vs. PD without FOG vs. matched controls; older adults vs. younger adults)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PD with FOG (Experimental): People with Parkinson's disease and freezing of gait:
  n = 25 in experiments 1 and 2, 20 in experiments 3 and 4. (Up to 90 participants, if each participant only volunteers for one study, however, the investigators anticipate a significant overlap and that most participants will volunteer for multiple experiments).
  Interventions: Device: EVS and EEG
- PD without FOG (Experimental): n = 25 in experiments 1 and 2, 20 in experiments 3 and 4. (Up to 90 participants, as in Group 1.)
  Interventions: Device: EVS and EEG
- Old adults matched controls (Active Comparator): (age- and sex-matched to the group with Parkinson's disease and freezing of gait): n = 25 in experiments 1 and 2, 20 in experiments 3 and 4. (Up to 90 participants, as in Group 1.)
  Interventions: Device: EVS and EEG
- young adults matched controls (Active Comparator): Young adults (age 21-44) n = 25 in experiments 1 and 2, 20 in experiments 3 and 4. (Up to 90 participants, as in Group 1.)
  Interventions: Device: EVS and EEG

INTERVENTIONS:
Device: EVS and EEG — The participant can choose to participate in one or more of the following experiments. (Any two of these visits will be separated by at least one week.) Experiment 1: EVS during gait initiation (forward stepping, 2 visits) Experiment 2: EVS during turning (1 visit) Experiment 3: EEG during gait initiation (forward stepping, 1 visit) Experiment 4: EEG during RAMS (1 visit)
  vestibular activity will be assessed using the noninvasive neuromodulation technique of electrical vestibular stimulation (EVS, Experiments 1 and 2) and cortical activity will be assessed by recording via electroencephalography (EEG, Experiments 3 and 4, no stimulation included).

SUMMARY:
Currently, there is a lack of comprehensive knowledge about the role of vestibulospinal drive and cortical activity during self-initiated movement transitions in older adults and people with PD (both with and without FOG). This set of experiments has two primary purposes: to (1) understand the pathological neurophysiology underlying freezing of gait (FOG) during movement transitions and FOG-inducing movements and (2) identify neurological biomarkers associated with FOG and FOG-inducing movements. To achieve this, the investigators will assess vestibular activity using the noninvasive neuromodulation technique of electrical vestibular stimulation (EVS, Experiments 1 and 2) and assess cortical activity by recording via electroencephalography (EEG, Experiments 3 and 4, no stimulation included). These experiments will investigate the vestibular (EVS Experiments) and cortical (EEG experiments) contributions to movement transitions during standing, walking, turning, and changing movement rates. Upon completion of this project, the investigators expect to provide a new understanding of key neural systems (vestibular and cortical) involved in the pathogenesis of movement impairment and freezing episodes during movement transitions including gait initiation, turning, and changing movement rates, in people with PD. An increased understanding of the temporal dynamics of systems involved in FOG and FOG-inducing movements could later guide the development and delivery of novel interventions (e.g. closed-loop deep brain stimulation [DBS] or non-invasive brain stimulation) to decrease the incidence and severity of FOG episodes, reducing fall risk and morbidity.

ELIGIBILITY:
Inclusion Criteria:

Participants with Parkinson's disease (with and without Freezing of Gait)

* Diagnosis of idiopathic PD.
* Age 40-80 years.
* Able to ambulate independently without the use of an assistive device (e.g. cane) for 50 meters. Healthy Older Adults (Control participants)
* Age 40-80 years (this group will be age- and sex-matched to the PD and FOG group).
* Able to ambulate independently without the use of an assistive device (cane or walker).
* Normal capacity to perform complex activities of daily living independently based on informant or physician report. Healthy Young Adults
* Age 21-44 years (this group will be sex-matched to the PD and FOG group)
* Able to ambulate independently without the use of an assistive device (cane or walker)

Exclusion Criteria:

Exclusion Criteria (for all participants):

* Any musculoskeletal disorder that affects the ability to stand or walk.
* History of musculoskeletal disorders that significantly affect movement of lower limbs.
* Uncorrected visual impairment that may affect participation or performance in the study.
* History of visual and/or vestibular conditions that may affect participation or performance in the study.
* Meet criteria for dementia with Lewy bodies, Multiple Systems Atrophy, Alzheimer's disease, dementia diagnosis, or other neurodegenerative disorder other than Parkinson's disease.
* History of seizures, epilepsy, stroke, multiple sclerosis, or traumatic brain injury or other significant neurological disorders that may affect participation or performance in the study.
* History of muscular conditions of the neck and back, including whiplash.
* History of surgery on blood vessels, brain, or heart.
* Unexplained, recurring headaches or concussion within the last six months.
* Moderate to severe hearing impairment.
* Subjects who are pregnant
* Reduced capacity to consent. This will be assessed using a 2-stage process. Initially, participants will be tested using the University of California, San Diego, Brief Assessment of Capacity to Consent (UBACC). If the results of the UBACC are inconclusive the individual will be further tested using the MacArthur Competency Assessment Tool for Clinical Research (McCAT-CR).

Additional exclusion criteria for EVS Experiments (Experiments 1 and 2):

* History of motion sickness (as EVS can exacerbate motion sickness).
* Intense physical exercise or consumption of alcohol in the 24 hours prior to any experiment that will include EVS testing.
* Recent history of migraine headaches.
* Intracranial metallic or magnetic devices.
* Pacemaker or any implanted device.
* Implanted deep brain stimulator or other neurosurgeries to treat PD.
* Use of medications that can cause dizziness.

Additional exclusion criteria for Control Participants:

* Presence of parkinsonism or cognitive impairment (including dementia or mild cognitive impairment).
* Active central nervous system, systemic, psychiatric conditions or use of psychoactive medication that would adversely affect cognitive, neuropsychiatric, motor, or autonomic functioning.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
timing of trunk muscle torque production | one day
  Onset and offset times of the trunk muscle activity, relative to the start of the turn, as measured by electromyography sensors
amplitude of trunk muscle torque production | one day
  Magnitudes of trunk muscle activity during the turn, as measured by electromyography sensors
ground reaction force | up to 3 days
  The forces resulting from the participant pushing into the floor during turns and gait initiation, as measured by force plates under the feet
center of pressure measures of turning and stepping | up to 3 days
  Participants will complete right/left 90 degree turns from standing on a pair of force plates (Kistler)
body segmental angular velocity | one day
  The speed at which different body parts (e.g., head, thoracic spine, etc.) rotate during a turn, as measured by 24 reflective markers at various bony landmarks on the head, trunk, pelvis, and lower extremities, used to capture the whole-body kinematic motion via optical motion capture various bony landmarks on their head, trunk, pelvis, and lower extremities to capture whole-body kinematic motion via optical motion capture (Simi Motion).
motion onset | up to 3 days
  Time of initial movement of the body, as measured by 24 reflective markers at various bony landmarks on the head, trunk, pelvis, and lower extremities, used to capture the whole-body kinematic motion via optical motion capture various bony landmarks on their head, trunk, pelvis, and lower extremities to capture whole-body kinematic motion via optical motion capture (Simi Motion).
total distance excursion | up to 3 days
  Distance moved, as measured by 24 reflective markers at various bony landmarks on the head, trunk, pelvis, and lower extremities, used to capture the whole-body kinematic motion via optical motion capture various bony landmarks on their head, trunk, pelvis, and lower extremities to capture whole-body kinematic motion via optical motion capture (Simi Motion).
Movement amplitude | one day
  Size of the movements, as measured by the manipulandum during repetitive movements
speed during the slow and fast epochs | one day
  Speed of the movements, as measured by the manipulandum during repetitive movements
duration of freezing events | one day
  Length of time during which movements are drastically decreased in size or speed nears zero, as measured by the manipulandum during repetitive movements
EVS coherence | up to 2 days
  1. A measure of the correlation between electrically evoked vestibular stimulation and the subsequent motor responses in the trunk and leg muscles prior to initiation of forward stepping or turning
  2. Coherence between trunk or leg muscle activation and EVS, coherence between ground reaction forces and EVS electrically evoked vestibular stimulation and the subsequent motor responses in the trunk and leg muscles prior to initiation of forward stepping
  coherence between trunk/leg muscle activation and EVS, coherence between ground reaction forces and EVS.

CONTACTS AND LOCATIONS:
Overall Officials: Sommer Huffmaster, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Movement Disorders Lab, Minneapolis, Minnesota, United States